CLINICAL TRIAL: NCT07360327
Title: Role of Opioid Free Anaesthesia in Elderly Patients Undergoing Elective Coronary Artery Bypass Graft Surgeries With Cardiopulmonary Bypass in Enhanced Recovery After Surgeries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: FMASU MD239/2025
Record Dates: First submitted 2025-12-05; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-10

CONDITIONS: CABG; Dexmedetomidine; Ketamine; Opioid Free Anesthesia; Opioid Based Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid free anesthesia group (Active Comparator): Patients will receive dexmedetomidine and ketamine
  Interventions: Drug: Opioid free anesthesia
- Opioid based group (Active Comparator): Patients will receive fentanyl
  Interventions: Drug: Opioid based Anesthesia

INTERVENTIONS:
Drug: Opioid free anesthesia — group (F) receive dexmedetomidine and ketamine
  Arms: Opioid free anesthesia group
Drug: Opioid based Anesthesia — Opioid based group receive fentanyl
  Arms: Opioid based group

SUMMARY:
The introduction of synthetic opioids in 1960 to general anesthesia together with sedative hypnotics and muscle relaxants allowed the appearance of the concept of multimodal balanced anesthesia. Although they help in achieving hemodynamic stability during anesthesia of open heart surgeries, their administration consequences are neither scarce nor benign to the patient. Perioperative opioids are associated with increased incidence of respiratory depression, prolonged mechanical ventilation, nausea and vomiting, prolonged sedation, Postoperative ileus (POI), urine retention, Postoperative cognitive dysfunction (POCD), immune depression and hyperalgesia (Beloeil et al., 2018).

Coronary artery bypass graft surgery with cardiopulmonary bypass (CPB) is particularly vulnerable to the above-mentioned complications. Indeed, some of the side effects of this surgery overlap with the adverse effects of opioids. Postoperative pulmonary complications are observed in up to 50% of patients (Fisscher et al., 2022) and POCD or delirium in 4-54% according to studies (Bhushan et al., 2021). Whereas major gastrointestinal complications are estimated to occur in around 3% of patients, essentially acute pancreatitis, postoperative ileus (Marsoner et al., 2019).

Opioid-free anesthesia (OFA) strategies have emerged to avoid intraoperative opioid use. It is based on the fact that a sympathetic reaction evidenced by hemodynamic changes in an anesthetised patient does not systematically reflect pain. In addition, a sleeping patient will not recall pain, while hormonal stress and sympathetic and inflammatory reactions can be controlled by therapeutic classes

DETAILED DESCRIPTION:
Study Procedures: o Randomization will allocate patients into two groups: Opioid-free (F) and Opioid-based (O) anesthesia, with numbers drawn from sealed envelopes. o Group F will receive analgesia through ketamine and dexmedetomidine based on Ideal Body Weight (IBW). o Group O will receive fentanyl for analgesia, also based on IBW. o IBW is calculated using ARDSnet formulas (Brower et al., 2000). o For men, IBW is 50 + (0.91 × [height in cm - 152.4]). o For women, IBW is 45.5 + (0.91 × [height in cm - 152.4]). o Patients will be monitored with ECG, pulse oximeter, and blood pressure monitoring before receiving midazolam for sedation. o After catheter insertion, patients will be assigned to groups based on the analgesia provided. o The analgesia will be prepared in a pharmacy, coded for blinding the anaesthetist. Fentanyl will be administered as follows: 3 mg/kg (IBW) for induction and 5 mg/kg for infusion during surgery (Baerdemaeker et al., 2004). • Ketamine and dexmedetomidine will be combined in one syringe with specific dosages for induction and infusion (Mulier et al., 2018). o Both groups will receive general anesthesia induction with midazolam, group-specific analgesia, propofol, and rocuronium before intubation. o Anesthesia maintenance will include isoflurane, group-specific analgesia infusion, and rocuronium infusions (Basagan et al., 2010).Hemodynamic parameters will be recorded at various intervals before and after induction until the patient is transferred to ICU. A 5mg bolus from the analgesia syringe will be administered for persistent tachycardia or hypertension, with a maximum of three doses before switching to second-line treatments. Norepinephrine will be given for significant hypotension. Propranolol will be administered for persistent tachycardia. Nitroglycerin will be used for persistent hypertension. Atropine will be given for severe bradycardia. Bradycardia, tachycardia, hypotension, and hypertension are defined based on specific heart rate and blood pressure changes. Propofol infusion will commence while on bypass and stop after weaning. Analgesia infusion will cease after sternum closure. Inhalational anesthetics will be discontinued at the end of the surgery, and patients will be transferred intubated and ventilated to ICU. In ICU, patients will be extubated once they meet specific requirements. Each group will be monitored for extubation timing and incidence of POCD using CAM ICU score. Cortisol levels and neutrophil lymphocytic ratio will be measured postoperatively in ICU. Patients will be excluded from the study for specific complications or delays. Post-operative analgesia will be administered regularly with paracetamol and fentanyl infusion or other analgesia in the respective groups.

ELIGIBILITY:
Inclusion Criteria:

* Age group: above 65 years old of both sex. Undergoing an elective coronary artery bypass graft surgeries with cardiopulmonary bypass.

Exclusion Criteria:

* Past or ongoing history of drug abuse.
* Psychiatric disease and cognitive disorders.
* Inability to perform the confusion assessment method for the intensive care unit (CAM-ICU) test.
* EF<40 %.
* 1st or 2nd degree Heart block.
* HR <50 bpm.
* Allergy from drugs used in this study.
* Use of a left ventricular assist device, IAB or ECMO pri

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Enhanced recovery time | 24 hours
  From transfer the patient to icu till extubation
Enhanced recovery defined as time of extubation | 24 hours
  Time from extubation after transfer to icu

SECONDARY OUTCOMES:
POCD | 1 week
  Post operative delerium by cam score which has 4 features ....to diagnose delerium patient must have 3 features
Post operative opioid consumption | IN the first 24 hour after surgery ...total morphine consumption
  Total morphine consumption
Cortisol level | 24 hours
  cortisol level